CLINICAL TRIAL: NCT04479683
Title: "COTIDEA COmparison Between Continued Inpatient Treatment Versus Day Patient Treatment (Partial Hospitalization) After Short Inpatient Care in Early Onset Anorexia Nervosa: a Non-inferiority Trial A Non-inferiority Study"
Brief Title: COmparison Between Continued Inpatient Treatment Versus Day Patient Treatment in Early Onset Anorexia Nervosa
Acronym: COTIDEA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP190069
Record Dates: First submitted 2020-07-08; First posted 2020-07-21 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Early Onset Anorexia Nervosa
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard care (Other): continuation of full-time hospitalization until the minimum healthy weight is reached, defined as the weight corresponding to the return to the previous BMI corridor (previous BMI +/- 1 BMI corridor, e.g. change from 25th to 10th percentile). This management combines bi-weekly medical follow-up by a senior psychiatrist, weekly family work, weekly therapeutic education group, weekly cognitive remediation group and bi-weekly dietary follow-up with therapeutic meals.
  Interventions: Other: standard care
- FTH (full-time hospitalisation) then day hospitalization) (Experimental): FTH output and DH relay one day a week until the minimum healthy weight. This treatment combines over one day a medical evaluation by a senior psychiatrist, family work (parents group and multi-family therapy session), a therapeutic education group, a cognitive remediation group and a dietary follow-up with therapeutic meals.
  During this phase, all children are evaluated once a week on a somatic level.
  Interventions: Other: FTH then DH support

INTERVENTIONS:
Other: FTH then DH support — FTH output and DH relay one day a week until the minimum healthy weight. This treatment combines over one day a medical evaluation by a senior psychiatrist, family work (parents group and multi-family therapy session), a therapeutic education group, a cognitive remediation group and a dietary follow-up with therapeutic meals.
  During this phase, all children are evaluated once a week on a somatic level.
  Arms: FTH (full-time hospitalisation) then day hospitalization)
Other: standard care — continuation of full-time hospitalization until the minimum healthy weight is reached, defined as the weight corresponding to the return to the previous BMI corridor (previous BMI +/- 1 BMI corridor, e.g. change from 25th to 10th percentile). This management combines bi-weekly medical follow-up by a senior psychiatrist, weekly family work, weekly therapeutic education group, weekly cognitive remediation group and bi-weekly dietary follow-up with therapeutic meals.
  Arms: standard care

SUMMARY:
"In so-called ""early onset"" anorexia nervosa (AN), a rare and severe form affecting 8-13 year olds, experts recommend that, as soon as possible, treatment should take place on an outpatient basis, at an age when separation from the usual environment would be particularly unpleasant and deleterious. However, in severe AN, full-time hospitalisation (FTH) is still indicated when somatic and psychiatric instability criteria are met. Thus, the severity and rapidity of undernutrition in children aged 8-13 years suffering from AN (linked on the one hand to the frequency of total aphagia with refusal to drink and on the other hand to the lack of early detection of the disorder, frequently requires emergency FTH, contrary to expert recommendations. This FTH, which lasts on average 3 months in our specialized unit, has certain disadvantages: poor acceptability by the patient and/or his family, increased anxiety symptoms on entry and exit, school dropout, social isolation, coercive experience. In addition, the rate of premature FTH exits - before weight targets are reached - and the frequency of relapses after FTH remain high, making FTH unsatisfactory in terms of cost-effectiveness. Some families refuse FTH, which is classically long, exposing themselves to the risk of complications that can occur if the disorder is inadequately treated: somatic, acute and chronic complications; risk of progression to another eating disorder.

In recent years, day hospitalization (DH) care has been developed for adolescents aged 11 to 18 years and adults (Madden, 2015). The few studies available are in favour of comparable efficacy, better acceptability and lower cost in the management of moderate AN compared to prolonged FTH, but also better social adaptation.In children aged 8 to 13 years with AN, whose somatic condition requires continuous monitoring in a hospital setting (the usual indication for FTH), a DH cannot reasonably be proposed immediately given the severity of the situation. Our hypothesis is that it would however be possible, in these children, to shorten the duration of FTH and to continue DH treatment once the critical period has passed at the somatic level, with comparable efficacy, best acceptability, best progress in terms of school and social integration, and lower cost.

DETAILED DESCRIPTION:
The objective of the study is to demonstrate the non-inferiority of DH management after a short full-time hospitalisation compared to a prolonged full-time hospitalisation aiming at a healthy weight on the evolution of BMI at 1 year in children aged 8 to 13 years suffering from anorexia nervosa, with severe undernutrition.

The minimum healthy weight is defined by a weight corresponding to the BMI corridor prior to the diagnosis of anorexia nervosa, +/- 1 corridor).

Randomized controlled trial, open-label, single-centre.

Patients will be randomized into one of the two arms of the trial:

* Group 1 (control group): continuation of full-time hospitalisation until reaching the minimum healthy weight, defined as the weight corresponding to the return to the previous BMI corridor (previous BMI +/- 1 BMI corridor, e.g. change from 25th to 10th percentile).
* Group 2 (experimental group): Exit from FTH (full-time hospitalisation ) and relay to DH (day hospitalization ) one day per week until the minimum healthy weight. This treatment combines a one-day medical evaluation by a senior psychiatrist, family sessions (parents group and multi-family therapy session), a therapeutic education group, a cognitive remediation group and a dietary follow-up with therapeutic meals.

Statistical analysis of the data will be carried out with the intention to treat. The BMI at 1 year between groups, as well as its bilateral 95% confidence interval (equivalent to a one-sided 97.5% confidence interval), will be estimated and compared with the predefined margin of non-inferiority (1 BMI point).

Ancillary study : Addition of a qualitative study conducted with parents to evaluate the implementation of a weekly intensive day hospital in the treatment of early-onset anorexia nervosa.

ELIGIBILITY:
Inclusion Criteria:

* Anorexia Nervosa according to diagnostic mental disorders(DSM 5) criteria;
* Age at diagnosis 8 to 13 years inclusive;
* Indication for full-time hospitalisation according to supreme health authority (HAS 2010) criteria, see appendix;
* First hospitalization in the Eating Disorders (ED) unit of the Child and Adolescent Psychiatry Department at Robert Debré Hospital.
* Informed consent of the holder(s) of parental authority
* Patient affiliated to a social security

Exclusion Criteria:

* Other early onset eating disorders (ARFID to DSM 5 criteria) ;
* Underlying unbalanced somatic disease (especially gastroenterological);
* Psychiatric indication for continued hospitalisation (in particular significant suicidal risk according to the psychiatric criteria for full-time hospitalisation for anorexia nervosa of the HAS, 2010, cf. appendix)
* Environmental indication for continued full-time hospitalization according to the HAS environmental criteria for full-time hospitalization for anorexia nervosa, 2010, cf. appendix) ;
* History of full-time hospitalisation in our ED unit.

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Estimated)
Dates: Start 2021-05-10 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
BMI BMI | one year
  body mass index (BMI) at 1 year after admission into FTH

SECONDARY OUTCOMES:
global clinical state | 3 months, 6 months and 1 year after admission into FTH
  Clinical global impression scale (CGI).Two "sub-scores": CGI-gravity and CGI-improvement.
  CGI-gravity measures the severity of a subject's current clinical condition (from 1 "normal, not at all sick" to 7 "among the sickest patients"). The improvement measures the perceived improvement in clinical status between assessments (rated from 1 "Very Much Improved" to 7 "Very Much Worsened").
Weight | at normalization of physiological parameters,3 months, 6 months and 1 year after admission into FTH
  Evaluate a healthy weight of a FTH intervention then DH versus conventional treatment
Height | at normalization of physiological parameters,3 months, 6 months and 1 year after admission into FTH
  Evaluate a height of a FTH intervention then DH versus conventional treatment
Number of weight recurrences | 12 months
  relapse risk assessment
number of rehospitalization days | 12 months
  relapse risk assessment
Quality of life of patients and parents | 6 months and 12 months
  Score on the satisfaction questionnaire (CSQ 8 and SF12)
Cost FTH then DH versus conventional treatment | 12 months
  Evaluate the efficiency of the FTH then DH versus FTH alone through a cost-utility analysis, and perform a cost-effectiveness analysis.
anxiety and depression | at normalization of physiological parameters,12 months
  The evolution of anxiety by Children Depression Inventory scale and State-Trait Anxiety Inventory
Self-esteem | at normalization of physiological parameters,12 months
  The evolution of self-esteem by Rosenberg self-esteem scale

CONTACTS AND LOCATIONS:
Overall Officials: Stordeur Coline, MD, Principal Investigator — APHP
Locations (1):
- Hôpital Robert Debré, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ayrolles A, Bargiacchi A, Clarke J, Michel M, Baillin F, Trebossen V, Kalifa HP, Guilmin-Crepon S, Delorme R, Godart N, Stordeur C. Comparison between continued inpatient treatment versus day patient treatment after short inpatient care in early onset anorexia nervosa (COTIDEA trial): a study protocol for a non-inferiority randomised controlled trial. BMC Psychiatry. 2023 Oct 10;23(1):730. doi: 10.1186/s12888-023-05222-9. PMID 37817147